CLINICAL TRIAL: NCT06063161
Title: Music Therapy for Hospitalized Patients With Parkinson's Disease and Lewy Body Dementia: A Randomized Controlled Pilot Trial to Prevent Delirium
Brief Title: Music Therapy to Prevent Hospital-acquired Delirium in Parkinson's Disease and Dementia With Lewy Bodies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Kara Smith, Associate Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H00001398
Record Dates: First submitted 2023-09-26; First posted 2023-10-02 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease; Dementia, Lewy Body; Delirium
Keywords: music therapy; music based intervention
MeSH Terms: conditions — Parkinson Disease; Lewy Body Disease; Delirium | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A blinded study coordinator will assess the primary outcome (Confusion Assessment Measure) to reduce bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy (Experimental): Music therapy intervention will be administered for 30 minutes 3 times per week between Day 0 and Day 15 of inpatient hospitalization. Daily passive music listening will be required for 30 minutes twice a day, at least 4 days per week. This daily listening experience will consist of personalized playlists developed by the music therapist with specific purpose and goal.
  Interventions: Behavioral: Music therapy intervention
- Standard care (Placebo Comparator): Usual standard care.
  Interventions: Other: Standard Care (in control arm)

INTERVENTIONS:
Behavioral: Music therapy intervention — Music therapy intervention administered for 30 minutes 3x/week by certified music therapist.
  Arms: Music Therapy
Other: Standard Care (in control arm) — placebo arm, routine standard care
  Arms: Standard care

SUMMARY:
The goal of this clinical trial is to test whether a music therapy intervention (MT) prevents hospital-acquired delirium (HaD) in patients with Parkinson's disease (PD) and Dementia with Lewy Bodies (DLB). Delirium is defined as a mental state in which you are confused, disoriented, and not able to think or remember clearly. It can start suddenly and is usually temporary. It is common among patients with PD/DLB during hospitalization.

We are conducting a randomized controlled feasibility pilot study of music therapy (MT) in patients with PD/DLB in the inpatient acute hospital setting.

We are testing if receiving music therapy lowers the risk of delirium, compared to other interventions. We are also testing if music therapy lowers the need for certain restraints and medications during the hospitalization.

Participants admitted to UMass Memorial Medical Center will be invited to participate. Participants will be asked to undergo a music therapy intervention for 30 minutes 3 times per week, and to listen to personalized music playlists for 60 minutes 4 times per week. Participants will be assessed for HaD every 24 hours, and will undergo additional surveys and questionnaires.

Researchers will compare the music therapy intervention to two another comparison groups: one group assigned to listen to music on their own, and one group assigned to receive only standard treatments. About one-third of the participants will be assigned to each of the three study groups.

DETAILED DESCRIPTION:
Participants will be screened within 24 hours of inpatient admission to UMass Memorial Medical Center, University Campus (Worcester, MA).

Participants will be randomized equally to one of three groups: 1) Music therapy (MT), 2) Active Control, 3) Standard of Care.

Participants will receive the assigned intervention within 48 hours of admission, and this will continue up to the day of discharge. If a participant remains hospitalized for more than 15 days, the assigned intervention will stop at Day 15.

The study groups are described below:

MT arm:

Participants will undergo one-on-one music therapy sessions of approximately 30 minutes duration, beginning within 48 hours of admission. Sessions will occur 3 times/week. Sessions will be conducted by a board-certified music therapist. Sessions will be customized to address patient needs but will consistently adhere to the four principal MT methods of re-creation, composition, improvisation, and therapeutic listening experiences. Sessions will be responsive to patient preferences, culture, and identity.

A research assistant will supervise and document details of each session on a validated intervention log, for instance time spent on each MT method, type of music utilized, and whether family was involved.

Participants will also receive a music "booster" of daily playlist listening. Developed by the music therapist, two 30-minute personalized playlists will be created taking into consideration the individual's preferences and level of function and cognition. One playlist will be developed to up-regulate alertness to improve orientation and participation in therapies and interventions, and a second playlist will be designed to down-regulate for relaxation/sleep and decreasing agitation. Playlists will be played for 30 minutes each daily (60 minutes total/day) using an iPad and either a speaker or noise cancelling headphones (depending on patient preference and music therapist recommendations) provided by the study team.

At study completion (date of discharge or Day 15 of hospitalization) +/- 2 days we will conduct semi-structured interviews with participants who received MT, and/or healthcare proxy/LAR, to understand perceptions of the MT program.

Active Control arm:

Those assigned to the active control arm will listen to music playlists for 30 min twice a day (1 hr total/day) 3x/week. Playlists will be generated automatically based on popular genres and not personalized. Participants will listen on an iPad using either a speaker or noise cancelling headphones (depending on patient preference and music therapist recommendations).Listening sessions will continue up to Day 15 of admission or until patient is discharged. During this time, routine orders for music therapy consults will not be allowed as part of usual inpatient care.

The rationale is to evaluate the differential impact of the one-on-one interaction with a music therapist compared to simple exposure to the music itself.

Standard of care (SoC) arm:

The SoC arm will receive the usual standard of care until discharge or Day 15 of hospitalization. During this time, routine orders for music therapy consults will not be allowed as part of usual inpatient care.

ELIGIBILITY:
Inclusion Criteria:

* Admitted as inpatient to UMass Memorial Medical Center University Campus
* Diagnosis of PD or DLB (ICD-10 G20 and G31.83 respectively) on active problem list or past medical history OR carbidopa/levodopa on active medication list or ordered in admission orders.

Exclusion Criteria:

* Severe hearing loss (unable to perceive sound < 71dB)
* Professed dislike or lack of reward with experiencing of all types of music (Barcelona Music Reward Questionnaire total score <40)
* History of musicogenic seizures
* Delirium present at initial assessment, as determined by a positive Confusion Assessment Method (CAM)
* Admitted to observation status or to Clinical Decision Unit (as these patients would not be expected to remain inpatient long enough to undergo the MT intervention)
* Patients who are currently prisoners will not be included
* Patients admitted and discharged within 24 hours.
* Patients in the intensive care unit receiving continuous intravenous sedative medication (as they would not be expected to be able to meaningfully participate in the study activities).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Confusion Assessment Measure (CAM) | administered at enrollment and once every 24 hours during study period
  A brief screening tool to assess for presence or absence of delirium

SECONDARY OUTCOMES:
Medication Administration Records and Orders | From enrollment up to 30 days after enrollment.
  We will measure recorded use and dosage of medications used to treat delirium. We will collect data on use of physical restraints and one-to-one sitters.

CONTACTS AND LOCATIONS:
Locations (1):
- UMass Medical School/UMass Memorial Medical Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
will be considered case by case by study team